CLINICAL TRIAL: NCT03317808
Title: Heavy Slow Resistance Exercise for Subacromial Pain Syndrome
Brief Title: Exercise for Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Hans-Hugo Fredriksen Høiland, Stud.med, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/1277
Record Dates: First submitted 2017-10-15; First posted 2017-10-23 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Subacromial Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy slow resistance exercise (Active Comparator)
  Interventions: Diagnostic Test: Different exercise
- Traditional supervised exercise (Placebo Comparator)
  Interventions: Diagnostic Test: Different exercise

INTERVENTIONS:
Diagnostic Test: Different exercise — Evaluating the difference between Heavy slow resistance and traditional exercise, based on the SPADI score.

SUMMARY:
This study evaluates the effect of Heavy Slow Resistance exercise (HSR) exercise in comparison with traditional supervised exercise as treatment for patients with subacromial shoulder pain. The purpose is to evaluate if HSR is feasible fir these patients, and compare its effect to traditional exercise at pain and function of the shoulder. One half will complete the heavy slow resistance exercise, the other will complete the conventional exercise.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain > Three months
* Subacromial pain
* Dysfunction or pain during abduction
* Pain during isometric strength test of abduction or external rotation of the shoulder.
* Positive Hawkins test
* Normal passive range of movement in the glenohumeral joint

Exclusion Criteria:

* Surgery of the affected shoulder
* Patients that are not considered suitable to complete the treatment, or able to answer a Norwegian questionnaire
* Shoulder dislocation or shoulder instability
* Clinical sign of cervical nerve root affection
* Rheumatoid arthritis
* Clinical sign of full rupture of the rotator cuff.
* Pregnancy
* Cortisone injection past six weeks

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline SPADI score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. Both dimensions account for 50% of the overall score, and scores from 0 to 100.

SECONDARY OUTCOMES:
Change from Baseline "Pain in rest last week" score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  11 point Likert-type scale, 0 =no pain, 10 = worst possible pain. Measured by marking a clean visual analogue scale, and later transferred to a score.
Change from Baseline "Pain in activity last week" score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  11 point Likert-type scale, 0 =no pain, 10 = worst possible pain. Measured by marking a clean visual analogue scale, and later transferred to a score.
Change From Baseline "The ability to carry a 5kg carry bag" score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  11 point Likert-type scale, 0 = no problem, 10 = impossible. Measured by marking a clean visual analogue scale, and later transferred to a score.
Change from Baseline DASH score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  DISABILITIES OF THE ARM, SHOULDER AND HAND (DASH) is a 30 points questionnaire about the disability of the shoulder. Answers from 0 to 5; 0 0 No problem completing the activity, 5 = Impossible to complete the activity. Total score is calculated by a summary of the scores, subtracted by 30 and divided by 1.2.
Change from Baseline Active range of motion of the shoulder at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  A total score the flection, abduction and external rotation of the shoulder. Measured by goniometer.
Change from "The ability to take something down from a high shelf" score at 12- and 24 weeks. | Measured three times. Firstly at the baseline. Secondly at the 12-week follow up (after finished intervention). Lastly at the 24-week follow up.
  11 point Likert-type scale, 0 = no problem, 10 = impossible. Measured by marking a clean visual analogue scale, and later transferred to a score.

CONTACTS AND LOCATIONS:
Overall Officials: Høiland, Principal Investigator — Oslo University Hospital
Locations (1):
- Ullevål Sykehus, Oslo, Norway